CLINICAL TRIAL: NCT01608906
Title: Efficacy of Low Dose Intravenous Heparin in Preventing Thromboembolism in the SICU.
Brief Title: Using Intravenous Heparin Versus Standard of Care Subcutaneous Heparin to Prevent Clots After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06-0854
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Results first posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Venous Thrombosis
Keywords: venous thrombosis; heparin; pulmonary embolism; ICU
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- continuous low dose intravenous heparin infusion (Experimental): titrated to a PTT of 40-45
  Interventions: Drug: low dose intravenous heparin (LDIVH)
- subcutanous heparin 5000 units 3 times/day (Active Comparator): standard of care
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: low dose intravenous heparin (LDIVH) — The LDIVH (experimental) group will receive a continuous heparin drip titrated to a prothrombin time (PTT) of 40-45. LDIVH subjects will have PTT tested within 24 hours prior to initiation of LDIVH. In addition, these subjects would continue to have a PTT tested every 6 hours until the PTT value falls between 40-45. All LDIVH subjects will have PTT values measured at least daily. This will continue until ICU discharge or a maximum of 28 days.
  Arms: continuous low dose intravenous heparin infusion
Drug: Heparin — 5000 units given subcutaneously three times a day until ICU discharge or a maximum of 28 days
  Arms: subcutanous heparin 5000 units 3 times/day

SUMMARY:
This study plans to learn more about what is the best treatment to prevent blood clots in patients in intensive care units (ICU's). The investigators know that patients who are in ICU's have a higher than normal risk of getting blood clots in the veins of their arms or legs. This can be very dangerous as the clot may move into the lungs. To prevent this, the standard treatment is to give low dose heparin subcutaneously 3 times a day (usually 5000 units at each dose). In this study the investigators are randomizing patients to receive either standard of care or low dose intravenous heparin in a continuous infusion.

DETAILED DESCRIPTION:
Macro- and micro-thrombosis both contribute significantly to morbidity and mortality in the surgical intensive care unit. Pulmonary embolism (PE) is a common and preventable cause of death in critically ill patients, with a mortality rate of up to 10%. Up to 95% of cases of PE originate from deep venous thrombosis (DVT). There are multiple pharmacologic and non-pharmacologic methods of DVT prophylaxis.The current standard of care in thromboprophylaxis in the surgical intensive care unit (SICU) at the University of Colorado Hospital is low-dose subcutaneous heparin (SCH). However, there is little evidence that this is the optimal prophylactic treatment. In fact, a database search of ICD-9 diagnoses made in 2005 suggests that the incidence of DVT in SICU patients, the majority who receive subcutaneous heparin, is approximately 7%. Surgical ICU patients are at high risk of developing DVT during their hospital stay and likely need more aggressive anticoagulation. Intravenous heparin, given at a low dose and titrated to a measurable endpoint PTT (partial thromboplastin time), may offer several benefits over the current standard of care, subcutaneous heparin. This method of treatment would offer more aggressive anticoagulation and allow dosage to be adjusted frequently based on each patient's changing coagulation status.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent;
* Age between 18 and 80 years
* The patient is admitted to the surgical intensive care unit at the University of Colorado Hospital

Exclusion Criteria:

* Predicated SICU stay less than 5 days;
* Pregnancy;
* Breast feeding;
* Initial platelet count < 30,000;
* Currently eligible for treatment of thromboembolism;
* Prior organ transplant;
* Cardiopulmonary bypass within previous 30 days;
* Advanced directive precluding participation;
* Already receiving pharmacologic agent for DVT prophylaxis;
* Prior diagnosis of heparin-induced thrombocytopenia;
* Heparin allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2007-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Cheng, MD; PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PI left the university in 2013. Numerous attempts were made to contact the PI and study team members, but efforts were unsuccessful. Arms are combined because no data is available regarding how participants were assigned to each study arm.
Groups:
- All Participants: Treatment: titrated to a PTT of 40-45. low dose intravenous heparin (LDIVH): The LDIVH (experimental) group will receive a continuous heparin drip titrated to a prothrombin time (PTT) of 40-45. LDIVH subjects will have PTT tested within 24 hours prior to initiation of LDIVH. In addition, these subjects would continue to have a PTT tested every 6 hours until the PTT value falls between 40-45. All LDIVH subjects will have PTT values measured at least daily. This will continue until ICU discharge or a maximum of 28 days.
  Control: Standard of Care.
Period: Overall Study
Arm/Group | All Participants
Started | 152
Completed | 113
Not Completed | 39

BASELINE CHARACTERISTICS:
Population: PI left the university in 2013. Numerous attempts were made to contact the PI and study team members, but efforts were unsuccessful. Arms are combined because no data is available regarding how participants were assigned to each study arm.
Arm/Group | All Participants
Number analyzed (Participants) | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 152
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 84
Region of Enrollment [Number; unit: participants]
  United States | 152

OUTCOME MEASURES:

1. Primary Outcome: Development of DVT (Deep Vein Thrombosis)
Description: In the first 70 patients, screening for DVT by ultrasound will occur on study days 0 and 5. After day 5 and for all remaining subjects, DVT will be diagnosed according to standard of care by the attending physician. Incidences of new DVT will be recorded daily until the patient is discharged from the hospital, or for a maximum of 28 days. DVT diagnosis will also be collected at 6 months from the primary care physician's office or the patient's household.
Time Frame: from start of study intervention to 6 months
Population: PI left the university in 2013. Numerous attempts were made to contact the PI and study team members, but efforts were unsuccessful. No outcome measure data is available
Arm/Group | Continuous Low Dose Intravenous Heparin Infusion | Subcutanous Heparin 5000 Units 3 Times/Day
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Development of PE's; Sepsis
Description: Secondary endpoints to be monitored for a maximum of 28 days, include: (1) total number of patients not developing PE; (2) total number of patients not developing sepsis; and (3) total number of patients not developing catheter-associated sepsis.
Time Frame: up to 28 days post study intervention start
Population: as for outcome 1
Arm/Group | Continuous Low Dose Intravenous Heparin Infusion | Subcutanous Heparin 5000 Units 3 Times/Day
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months.
Description: PI left the university in 2013. Numerous attempts were made to contact the PI and study team members, but efforts were unsuccessful. Arms are combined because no data is available regarding how participants were assigned to each study arm.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/152
Serious Adverse Events (participants affected / at risk) | 0/152
Other Adverse Events (participants affected / at risk) | 0/152

LIMITATIONS AND CAVEATS:
PI left the university in 2013. Numerous attempts were made to contact the PI and study team members to obtain results data, but efforts were unsuccessful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No